CLINICAL TRIAL: NCT07230158
Title: The Effects of TRanscranial AlterNating Current Stimulation FOR Patients With Mild Alzheimer's Disease II (TRANSFORM-AD II Study): A Randomized Controlled Clinical Trial
Brief Title: Transcranial Alternating Current Stimulation for Patients With Mild Alzheimer's Disease II (TRANSFORM-AD II)
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Xuanwu Hospital, Beijing (Other)
Collaborators: Beijing Geriatric Hospital (Other); The First Affiliated Hospital of Zhengzhou University (Other); First Affiliated Hospital of Chongqing Medical University (Other); The Fifth People's Hospital of Datong (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2023173
Record Dates: First submitted 2025-09-21; First posted 2025-11-17 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Alzheimer Disease
MeSH Terms: conditions — Alzheimer Disease | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- tACS stimulation group (Experimental): NEXALIN ADI transcranial alternating current stimulator
  Interventions: Device: transcranial alternating current stimulation
- sham stimulation group (Sham Comparator): Sham stimulator provided by NEXALIN company
  Interventions: Device: sham stimulation

INTERVENTIONS:
Device: sham stimulation — Electrodes will also be placed on the patient's forehead and behind both ears. The sham stimulator is identical in appearance to the true stimulator. Neither participants nor operators can distinguish whether the stimulator is real based on its appearance or the patient's sensations. However, when the device is activated, no current flows through the electrodes. Participants in this group will receive sham stimulation with 60 one-hour sessions within 8 weeks.
  Arms: sham stimulation group
Device: transcranial alternating current stimulation — The alternating current is delivered through medical-grade conductive electrode pads manufactured specifically for Nexalin technology. The electrode pads are placed on the forehead and behind both ears, and are connected to the Nexalin device with thin cables. The intervention will be conducted with a tACS device: 50 minutes of high-gamma frequency (77.5 Hz) combined with 10 minutes of low-gamma frequency (40 Hz), with a peak-to-peak amplitude of 15 mA. A total of 60 one-hour sessions will be completed within 8 weeks.
  Arms: tACS stimulation group

SUMMARY:
The goal of this study is to explore the efficacy and safety of transcranial alternating current stimulation (tACS) in patients with amnestic mild cognitive impairment due to Alzheimer's disease (AD-aMCI) and patients with mild Alzheimer's disease dementia (AD-MD). The study will recruit 160 individuals with mild cognitive impairment with evidence of amyloid plaques in the brain through Positron Emission Tomography (PET) imaging. Participants will undergo baseline cognitive assessment, structural and functional MRI characterization, PiB-PET, and EEG measurement. The participants will be randomized to either a tACS group or a sham stimulation group. At the end of the intervention, all subjects will repeat the baseline assessments.

DETAILED DESCRIPTION:
Background In our previous study, we applied 40 Hz transcranial alternating current stimulation (tACS) to patients with mild Alzheimer's disease (AD), and the results demonstrated significant improvements in cognitive function. Building upon these findings, the present study applies a combined high-gamma (77.5 Hz) and low-gamma (40 Hz) tACS protocol to target patients with amnestic mild cognitive impairment due to Alzheimer's disease (AD-aMCI) and those with mild Alzheimer's disease dementia (AD-MD). This dual-frequency stimulation aims to enhance cognitive performance through synergistic gamma-band modulation and to explore its underlying therapeutic mechanisms.

Methods The TRANSFORM-AD II trial is a double-blind, randomized controlled study that will enroll 160 participants diagnosed with AD-aMCI or AD-MD. Eligible participants must meet at least one of the following criteria: positive amyloid positron emission tomography (PET), decreased cerebrospinal fluid (CSF) amyloid-β levels, or elevated plasma phosphorylated tau 217 (p-Tau217) levels. Participants will be randomly assigned to either the active stimulation group (77.5 Hz + 40 Hz tACS) or the sham stimulation group. Both groups will receive 60 one-hour sessions over an 8-week period. Outcome measures will be assessed at baseline and immediately after the intervention.

The primary outcome is global cognitive function, measured using the Alzheimer's Disease Assessment Scale-Cognitive Subscale (ADAS-Cog 13).

Secondary outcomes include changes in other neuropsychological test scores, multimodal magnetic resonance imaging (MRI) metrics, and resting-state as well as task-related electroencephalography (EEG) indicators.

Results This trial is currently ongoing, with recruitment expected to be completed by June 2026.

Conclusion This study will evaluate the efficacy and safety of combined 77.5 Hz and 40 Hz tACS in patients with AD-related aMCI and mild AD dementia. Furthermore, it will investigate potential therapeutic mechanisms using multimodal MRI to assess brain structure and function, and EEG to characterize both resting-state and task-related neural activity patterns.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged 50-90 years, either inpatients or outpatients;
2. Meeting the NIA-AA clinical diagnostic criteria established by the 2018 National Institute on Aging and Alzheimer's Association (NIA-AA) group for AD-related amnestic mild cognitive impairment (a-MCI) or AD-related mild dementia;
3. Neuropsychological evaluation with MMSE score of 18-26 and CDR score of 0.5 or 1;
4. Positive amyloid PET, or decreased amyloid levels in cerebrospinal fluid, or elevated serum phosphorylated Tau217 protein;
5. Able to communicate proficiently in Chinese (non-illiterate);
6. If currently receiving cholinesterase inhibitor treatment (such as donepezil or rivastigmine), the current treatment dose must be stable (i.e., fixed dose for at least 6 consecutive weeks), with no planned dose adjustments during the study observation period;
7. Signed informed consent form.

Exclusion Criteria:

1. Sudden onset;
2. Early focal neurological manifestations or extrapyramidal manifestations;
3. Systemic diseases that may cause cognitive impairment (such as liver or kidney insufficiency, endocrine diseases, or vitamin deficiency), or neurological diseases such as brain trauma, epilepsy, encephalitis, or normal pressure hydrocephalus;
4. Meeting DSM-IV criteria for depression or schizophrenia;
5. Ongoing drug treatments that may affect baseline or follow-up assessments;
6. Contraindications for MRI or neurophysiological examinations, such as cardiac pacemakers, cardiac defibrillators, implanted electronic systems, vascular clips, mechanical heart valves, or cochlear implants;
7. Cranial MRI showing ischemic lesions meeting NINCDS-AIREN criteria.

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2025-11-30 (Estimated); Primary Completion 2027-09-01 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
Change in Alzheimer's Disease Assessment Scale cognitive subscale (ADAS-cog, 13-items version). | up to 8 weeks (end of intervention)
  ADAS-cog 13 scale ranges from 0 to 85, and higher value represents a worse outcome. This study will use ADAS-cog to assess changes in the global cognitive function after intervention.

SECONDARY OUTCOMES:
Change in MRI brain connectivity | up to 8 weeks (end of intervention)
  Functional MRI and DTI will be used to measure the connectivity of different ROIs, and the intervention effect will be evaluated by assessing changes in connectivity indicators before and after the intervention.
Temporal lobe cross-frequency coupling dynamics and intervention effects | Up to 8 weeks (end of intervention)
  This study aims to evaluate the dynamic changes in cross-frequency coupling (CFC) indices within the temporal lobe across different time points following intervention. By analyzing phase-amplitude coupling between distinct frequency bands, the study seeks to characterize alterations in α-γ and θ-γ coupling patterns in individuals with migraine and epilepsy. The findings will help elucidate the role of temporal lobe functional connectivity in disease progression and in the modulation of non-pain symptoms.
Changes in brain volume and brain function | up to 8 weeks (end of intervention)
  Structural and functional MRI will be used to measure brain structure and brain function
Change in Mini-mental State Examination | up to 8 weeks (end of intervention)
  Mini-mental State Examination (MMSE) will be used to evaluate the general cognitive function. MMSE ranges from 0 to 30, and higher value represents a better outcome.
Change in Montreal Cognitive Assessment | up to 8 weeks (end of intervention)
  Montreal Cognitive Assessment (MoCA) will be used to evaluate the general cognitive function. MoCA ranges from 0 to 30, and higher value represents a better outcome.
Change in Clinical Dementia Rating Scale sum of the boxes | up to 8 weeks (end of intervention)
  Clinical Dementia Rating Scale sum of the boxes (CDR-SB) will be used to evaluate the general cognitive function. CDR-SB ranges from 0 to 18, and higher value represents a worse outcome.
Change in memory function | up to 8 weeks (end of intervention)
  WHO-UCLA Auditory Verbal Learning Test will be used to assess memory function. It ranges from 0 to 45, and higher values represent better outcomes. In addition, task-related EEG will be conducted during memory tasks to further evaluate memory-related neural activity.
Change in Digit span forward | up to 8 weeks (end of intervention)
  Digit span will be used to assess attention. It ranges from 3 to 10, and higher value represents a better outcome.
Change in Digit span backward | up to 8 weeks (end of intervention)
  Digit span backward will be used to assess executive function. It ranges from 2 to 8, and higher value represents a better outcome.
Change in Trail Making Test | up to 8 weeks (end of intervention)
  Trail-Making Test B minus A score will be used to assess executive function. Trail-Making Test B minus A ranges from -150 to 300, higher value represents a worse outcome.
Change in Boston Naming Test | up to 8 weeks (end of intervention)
  Boston Naming Test will be used to assess language function. It ranges from 0 to 30, and higher value represents a better outcome.
Change in Neuropsychiatric Inventory (NPI) | up to 8 weeks (end of intervention)
  The Neuropsychiatric Inventory will be used to measure neuropsychiatric symptoms. It ranges from 0 to 144, and higher value represents a worse outcome.
Change in Geriatric Depression Scale (GDS) | up to 8 weeks (end of intervention)
  The Geriatric Depression Scale will be used to measure neuropsychiatric symptoms. It ranges from 0 to 30, and higher value represents a worse outcome.
Change in Activities of Daily Living | up to 8 weeks (end of intervention)
  Activities of Daily Living (ADL) scale will be used to assess the change of life quality. It ranges from 20 to 80. The "20" represents normal life ability and the higher score presents the worse life ability.
Side-effects of tACS | up to 8 weeks (end of intervention)
  Adverse Events as a result of tACS stimulation will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Yi Tang, M.D., Ph.D., Principal Investigator — Xuanwu Hospital, Beijing
Locations (1):
- Xuanwu Hospital, Capital Medical University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
Study Protocol, Statistical Analysis Plan (SAP), Informed Consent Form (ICF), Clinical Study Report (CSR), Analytic Code
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: 2025.9.20-2027.9.20